CLINICAL TRIAL: NCT00801736
Title: A Multicentre, Randomised, Phase III Trial of Platinum-based Chemotherapy Versus Non-platinum Chemotherapy, After ERCC1 Stratification, in Patients With Advanced/Metastatic Non-small Cell Lung Cancer
Brief Title: ERCC1 Targeted Trial
Acronym: ET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The antibody used did not appear prognostic/predictive based on interim results.
Sponsor: University College, London (Other)
Collaborators: Eli Lilly and Company (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN02370070; CRUK-UCL-ET; EUDRACT-2007-007639-17
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Lung Cancer
Keywords: Recurrent non-small cell lung cancer; Stage IIIB non-small cell lung cancer; Stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platinum Arm (Experimental): Cisplatin (IMP) / Pemetrexed (IMP)
  Interventions: Drug: Cisplatin, Paclitaxel
- Non Platinum Arm (Experimental): Paclitaxel (IMP) / Pemetrexed (IMP)
  Interventions: Drug: Cisplatin, Paclitaxel

INTERVENTIONS:
Drug: Cisplatin, Paclitaxel — * Cisplatin 75mg/m2, Day 1
  * Paclitaxel 175mg/m2, Day 1

SUMMARY:
Lung cancer is the leading cause of cancer death in the UK, leading to 34 000 deaths each year (22% of cancer deaths). Non-small cell lung cancer (NSCLC) is the most common histology, accounting for approximately 80% of cases and most present with advanced, stage IIIb or IV disease. The recommended treatment for advanced disease is a doublet platinum-based chemotherapy, although the survival benefits are modest. Even among those fit enough for chemotherapy, the response rate is only 20-40%, and median survival averages 9-10 months with the newer platinum-containing chemotherapy regimen (Schiller et al, 2002; Rudd et al, 2005; Lee et al, 2007). Only 11% of patients went on to survive 2 years when treated with the newer gemcitabine/carboplatin regimen established by the London Lung Cancer Group (Rudd et al, 2005; Lee et al, 2007). New strategies are needed to further improve the prognosis of this disease.

DETAILED DESCRIPTION:
TRIAL OBJECTIVES

Primary objective

The trial will have two main objectives:

* To detect an improvement in survival for ERCC1+ve patients treated with a non-platinum chemotherapy compared to platinum-based treatment.
* To establish non-inferiority or improvement in survival for ERCC1-ve patients treated with a platinum-based chemotherapy compared to non-platinum treatment.

Secondary objectives

* To examine progression-free survival, response rate and quality of life between the two treatment regimens, according to ERCC1 status.
* To investigate whether the treatment effect differs according to histology (squamous vs. nonsquamous);gender (males vs. females); performance status
* To undertake a cost-effectiveness analysis based on all patients, and according to ERCC1 status.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histological confirmation of non-squamous NSCLC
2. Have a tissue biopsy available for sending to the central laboratory to determine ERCC1 status
3. Presentation with stage IIIb (not amenable to curative treatment) or IV disease - staging scans must be no more than 28 days prior to registration. Patients with relapsed NSCLC must not have received prior chemotherapy or biological therapy (previous surgery or radical radiotherapy allowed)
4. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours
5. Either sex, at least 18 years of age
6. ECOG performance status 0-1
7. Estimated life expectancy of at least 8 weeks
8. Adequate bone marrow function as evidenced by the following (assessed within 14 days of registration):

   * Absolute neutrophil count (ANC) ≥1.5 × 109/L
   * Platelet count ≥100 × 109/L
   * Haemoglobin ≥9 g/dL
9. Adequate liver function as evidenced by the following (assessed within 14 days of registration):

   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) ≤3 × ULN or ≤5 × ULN is acceptable with liver metastases
   * Alanine transaminase (ALT) ≤3 × ULN
10. Adequate renal function as evidenced by the following (assessed within 14 days of registration):

    - GFR > 60ml/min as measured by creatinine clearance through EDTA. Alternatively, the Cockcroft and Gault formula may be used to estimate GFR, but if < 60 ml/min then EDTA should be performed.
11. Previous palliative radiotherapy to non-target metastatic lesions is allowed for pain relief prior to starting chemotherapy
12. Patients with stable brain metastases will be allowed to enrol. Stable brain metastases being defined as no progression of brain metastases 28 days after treatment as documented by a CT scan/MRI of the brain. Patients with incidentally discovered asymptomatic brain metastases may be enrolled and treated with trial chemotherapy without prior brain irradiation if deemed feasible by the treating physician
13. Signed informed consent form
14. Use of effective contraception during, and for 6 months after trial treatment by patients of reproductive potential and partners of reproductive potential. Patients who receive aprepitant (anti-emetic) must be willing to use an alternative or back-up method to hormonal contraceptives as aprepitant may reduce their efficacy. Female patients with childbearing potential must have a negative serum pregnancy test prior to registration.

EXCLUSION CRITERIA

1. Cytologically or clinically diagnosed NSCLC
2. Evidence of significant medical condition or laboratory finding which, in the opinion of the treating physician or chief investigator, makes it undesirable for the patient to participate in the trial
3. Presence of uncontrolled brain or leptomeningeal metastases thought to require immediate radiotherapy
4. Presence of clinically significant third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to trial entry
5. Yellow fever vaccination received within the 30 days previous to study entry
6. Unable to interrupt aspirin or other NSAIDs (for pemetrexed arms of the trial)
7. Unable or unwilling to take vitamin B12 and folic acid (for pemetrexed arms of the trial)
8. A history of prior malignant tumour, unless the patient has been without evidence of disease for at least 3 years or the tumour was a non-melanoma skin tumour or early cervical cancer
9. Pregnant or lactating women
10. Inability to comply with protocol or trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Dec 2014

SECONDARY OUTCOMES:
Time to progression | Dec 2014

CONTACTS AND LOCATIONS:
Overall Officials: Siow M. Lee, MD, PhD, FRCP, Principal Investigator — Cancer Research UK
Locations (1):
- University College London Hospitals, London, United Kingdom